CLINICAL TRIAL: NCT02674763
Title: A Phase 1, Multi-center, Open-label Study of IMGN779 Administered Intravenously in Adult Patients With Relapsed/Refractory CD33-positive Acute Myeloid Leukemia
Brief Title: Open-label Study of IMGN779 in Adult Patients With Relapsed/Refractory CD33-positive Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ImmunoGen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMGN779 0601
Record Dates: First submitted 2016-02-01; First posted 2016-02-04 (Estimated); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; AML; IMGN779; ImmunoGen; Phase 1; Relapsed; Refractory; CD33; Dose Escalation; Dose Expansion
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Dose Escalation Schedule A (Experimental): IMGN779 administered on days 1 and 15 of a 28-day cycle
  Interventions: Drug: IMGN779
- Dose Escalation Schedule B (Experimental): IMGN779 administered on days 1, 8, 15 and 22 of a 28-day cycle
  Interventions: Drug: IMGN779
- Dose Escalation Schedule C (Experimental): IMGN779 administered on days 1 and 8 of a 21-day cycle
  Interventions: Drug: IMGN779
- Dose Expansion Cohort (Experimental): Patients with Relapsed AML; IMGN779 administered at dose and schedule selected as the putative RP2D.
  Interventions: Drug: IMGN779

INTERVENTIONS:
Drug: IMGN779

SUMMARY:
This is an open label, multicenter Phase 1 study to determine the MTD, dosing schedule and RP2D of IMGN779 when administered as mono-therapy to adult AML patients with CD33 -positive disease.

DETAILED DESCRIPTION:
In the Dose Escalation Phase, patients will be assigned to one of three schedules. The MTD for all schedules will be determined from the assessment of Dose Limiting Toxicities (DLTs). The Dose Expansion Phase will consist of one cohort based on patients response to prior therapy according to the MTD selected.

ELIGIBILITY:
Inclusion Criteria:

* Dose Escalation: Patients with relapsed or refractory AML
* Dose Expansion: Patients with relapsed AML or patients who refuse, or are not suitable candidates for induction therapy

Exclusion Criteria:

* Dose Escalation: Acute Promyelocytic Leukemia
* Any concurrent anti-cancer therapy including chemotherapy, immunotherapy, radiotherapy, biologic or any investigational agents (with the exception of hydroxyurea or leukapheresis for control of hyperleukocytosis) within 14 days or five half-lives of drugs, whichever is shorter, prior to Cycle 1 Day 1
* AML patients with known, active leptomeningeal/central nervous system (CNS) involvement
* Prior treatment with IMGN779
* Women who are pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of IMGN779 | 28 days

SECONDARY OUTCOMES:
Treatment emergent adverse events | Up to 12 months
Objective Response Rate (ORR) (complete response [CR= CR+CRp+CRi]+partial remission [PR]) | Up to 12 months
PK parameters: maximum plasma concentration (Cmax) of IMGN779 | up to 12 months
PK parameters: area under the time-concentration curve (AUC) of IMGN779 | Up to 12 months
PK parameters: terminal half-life (t½) of IMGN779 | Up to 12 months
Immunogenicity: Presence of Antibody-Drug Antibody (ADA) | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Zweidler-McKay, MD, Study Director — ImmunoGen, Inc.
Locations (7):
- United States (7):
  - Comprehensive Cancer Center (UAB CCC), Birmingham, Alabama
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - New Mexico Cancer Care Alliance, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Knight Cancer Institute - OSHU, Portland, Oregon
  - Baylor Scott & White University Medical Center, Dallas, Texas
  - The University of Texas, MD Anderson Cancer Center, Houston, Texas